CLINICAL TRIAL: NCT00683059
Title: A Multi-Institutional Phase II Study of Single Agent Abraxane as Second Line Therapy in Patients With Advanced Transitional Cell Carcinoma of the Urothelium
Brief Title: Single Agent Abraxane as Second Line Therapy in Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABX207-GU07CA
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Transitional Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nab-paclitaxel (Experimental)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — total dose (mg) = body surface area in m2 x study dose (mg/m2) to be injected into a vein once every 3 weeks over 18 months.
  Other Names: Abraxane

SUMMARY:
The purpose of this study is to determine what effects the drug Abraxane has on bladder cancer.

DETAILED DESCRIPTION:
For those patients with advanced bladder cancer who have progressed on a platinum based regimen, no widely accepted standard second line therapy currently exists. Taxanes including paclitaxel have exhibited clinical activity in this disease and are sometimes given off study. However, toxicities including neurotoxicity and hypersensitivity reactions often limit the use of paclitaxel. ABRAXANE may allow delivery of a greater dose of paclitaxel to those with bladder cancer with an easier method of administration and with less toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological or cytological diagnosis of urothelial carcinoma. Mixed histologies are permitted as long as transitional cell carcinoma is the major component (i.e. >50% of the pathologic specimen). Pure or predominant squamous cell carcinomas are not permitted.
* Patients with transitional cell carcinomas of the renal pelvis and ureter are permitted.
* Patients must have metastatic or locally advanced unresectable disease.
* Patients must have received one and only one prior chemotherapeutic regimen which included a platinum (at least one cycle) for metastatic/recurrent disease. Neoadjuvant or adjuvant chemotherapy will be considered to have been first line if the patient progressed within 12 months of the last dose.
* Neoadjuvant/adjuvant chemotherapy (with or without a taxane) is permitted if registration is greater than 12 months since the last dose (patients must then have received one platinum containing regimen in the metastatic setting)
* ECOG performance status <= 2.
* Estimated life expectancy of >12 weeks.
* Patients must have measurable disease according to RECIST criteria.
* If female of childbearing potential, pregnancy test is negative within 72 hours priors to first dose of study drug.
* If fertile, patient agrees to use an effective method of contraception to avoid pregnancy for the duration of the study.
* Adequate organ function; Absolute neutrophil count >1.5 x 109/L. Platelet count >100 x109/L. Hemoglobin >90 g/L. Total bilirubin <1.5x upper limit of normal. Transaminases <3x upper limit of normal (<5x if liver metastasis are present) Calculated creatinine clearance >40 ml/min (Cockcroft & Gault formula)
* Able to give informed consent.

Exclusion Criteria:

* Prior taxane therapy for metastatic disease (or > 12 months since a taxane-containing neoadjuvant or adjuvant chemotherapy).
* Pre-existing peripheral neuropathy >1 by NCI-CTC criteria.
* Pregnant or lactating females.
* Uncontrolled brain or leptomeningeal involvement (treated brain metastasis permitted if both known lesions and medications e.g. steroids for that indication are stable).
* History of serious or concurrent illness that might be aggravated by study treatment.
* History of class II-IV congestive heart failure.
* Other malignancies except adequately controlled basal cell carcinoma of the skin or carcinoma in situ of the cervix or incidental prostate cancer (T1a, Gleason <7 PSA <10ng/ml) or any other tumor within 5 years prior to enrollment.
* Other investigational therapy or radiation therapy within 30 days before registration.
* Patients not willing to employ adequate contraception for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Response rate | one year

SECONDARY OUTCOMES:
safety | 1 year
overall survival | 1-2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yoo-Joung Ko, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (5):
- Canada (5):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Ko YJ, Canil CM, Mukherjee SD, Winquist E, Elser C, Eisen A, Reaume MN, Zhang L, Sridhar SS. Nanoparticle albumin-bound paclitaxel for second-line treatment of metastatic urothelial carcinoma: a single group, multicentre, phase 2 study. Lancet Oncol. 2013 Jul;14(8):769-76. doi: 10.1016/S1470-2045(13)70162-1. Epub 2013 May 22. PMID 23706985